CLINICAL TRIAL: NCT02667041
Title: NeuroQore Repetitive Transcranial Magnetic Monophasic vs. Biphasic Stimulation For Major Depressive Disorder: A Randomized Controlled Trial
Brief Title: NeuroQore rTMS (Monophasic vs. Biphasic) for Major Depressive Disorder: A Randomized Controlled Pilot Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Collaborators: NeuroQore Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Verner Knott, Neuroelectrophysiology and Cognitive Research Laboratory, Director, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015014
Record Dates: First submitted 2016-01-25; First posted 2016-01-28 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- rTMS treatment (Monophasic vs. biphasic) (Experimental): Safety and efficacy
  Interventions: Device: NeuroQore rTMS Device
- EEG/ERP biomarkers (Active Comparator): Investigation of pre- and post-treatment cognitive biomarkers
  Interventions: Device: NeuroQore rTMS Device
- Blood biomarkers (Active Comparator): Investigation of pre- and post-treatment protein biomarkers
  Interventions: Device: NeuroQore rTMS Device

INTERVENTIONS:
Device: NeuroQore rTMS Device

SUMMARY:
Major depressive disorder (MDD) is a debilitating illness that affects millions of individuals in North America and can result in clinical symptoms including loss of pleasure and feelings of worthlessness, in addition to significant cognitive impairments (e.g., memory, attention) that affect daily functioning. Major depression bears a heavy burden for the individuals and family members afflicted, as well as an enormous health care and economic cost. Approximately half of major depressive patients seek out treatment for their illness and only 20% of those individuals report their treatment as satisfactory. Many MDD patients do not respond to pharmacological therapy following the first course of treatment, resulting in the need for alternative measures to alleviate the clinical and cognitive symptoms of treatment-resistant depression and the targeting of these therapies to better suit each individual patient. Repetitive transcranial magnetic stimulation (rTMS) is a well-accepted, non-invasive technique that utilizes currents to induce electrical fields that excite specific brain regions. The current recommended practice of rTMS involves the administration of a biphasic stimulus waveform; however, a novel method using monophasic pulses may prove more effective for the treatment of depression. The present study aims to determine the effect of monophasic rTMS compared to biphasic rTMS on cognitive processing in MDD patients through electrophysiological recordings of the brain taken before and after 6 weeks of stimulation. Additionally, the study aims to investigate various biological markers linked to clinical rTMS response; these brain markers will help in personalizing treatment for individuals suffering from MDD.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included if they:

1. are outpatients of the ROHCG
2. are voluntary and competent to consent to treatment
3. have a confirmed DSM-IV diagnosis of unipolar major depressive disorder
4. are male or female
5. are between the ages of 18 and 75
6. have failed to achieve a clinical response to an adequate dose of an antidepressant in the current episode OR have been unable to tolerate at least 2 separate trials of antidepressants of inadequate dose and duration
7. have a score > 22 on the MADRS
8. have had no increase or initiation of any psychotropic medication in the 4 weeks prior to screening
9. are able to adhere to the treatment schedule
10. pass the TMS safety screening questionnaire (TASS)
11. have normal thyroid functioning based on pre-study blood work

Exclusion Criteria:

Patients will be excluded if they:

1. have a history of substance dependence or abuse within the last 3 months or current substance use as indicated by a positive urine drug screen
2. have a concomitant major unstable medical illness, cardiac pacemaker or implanted medication pump
3. have active suicidal intent
4. are pregnant
5. have a lifetime DSM-IV diagnosis of bipolar I or II disorder, schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, or current psychotic symptoms
6. have a DSM-IV diagnosis of obsessive compulsive disorder, post-traumatic stress disorder (current or within the last year), anxiety disorder (generalized anxiety disorder, social anxiety disorder, panic disorder), or dysthymia, or personality disorder, assessed by a study investigator to be primary and causing greater impairment than MDD
7. have failed a course of ECT in the current episode or previous episode
8. have received rTMS for any previous indication due to the potential compromise of subject blinding
9. have any significant neurological disorder or insult including, but not limited to: any condition likely to be associated with increased intracranial pressure, space occupying brain lesion, any history of seizure except those therapeutically induced by ECT, cerebral aneurysm, Parkinson's disease, Huntington's chorea, multiple sclerosis, significant head trauma with loss of consciousness for greater than or equal to 5 minutes
10. have an intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed
11. if participating in psychotherapy, must have been in stable treatment for at least 3 months prior to entry into the study, with no anticipation of change in the frequency of therapeutic sessions, or the therapeutic focus over the duration of the study
12. clinically significant laboratory abnormality, in the opinion of the investigator
13. currently (or in the last 4 weeks) take more than lorazepam 2 mg daily (or equivalent) or any dose of an anticonvulsant due to the potential to limit rTMS efficacy
14. non-correctable clinically significant sensory impairment (i.e., cannot hear well enough to cooperate with interview)
15. failure of 3 or more adequate trials of medications of different drug classifications in the current episode

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-05; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) scores | Six weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Ottawa Mental Health Centre, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Goodman MS, Blumberger DM, Talebinejad M, Chan ADC, Chen R, Yang TT. Rectangular Repetitive Transcranial Magnetic Monophasic vs Biphasic Stimulation for Major Depressive Disorder: A Randomized Controlled Pilot Trial. Neuromodulation. 2025 Apr;28(3):511-519. doi: 10.1016/j.neurom.2024.11.010. Epub 2025 Jan 6. PMID 39772341